CLINICAL TRIAL: NCT02727452
Title: Effects of Immediate Bonding (Skin-to-skin Contact) During Caesarean Section- Psychobiological and Somatic Outcomes of Mother and Child
Brief Title: Immediate Bonding and Caesarean Section
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johann Wolfgang Goethe University Hospital (Other)
Responsible Party: Principal Investigator, Dr. Silvia Oddo, Dr.rer.nat., Johann Wolfgang Goethe University Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: E 9/15
Record Dates: First submitted 2015-10-12; First posted 2016-04-04 (Estimated); Last update posted 2022-03-15 (Actual); Status verified 2022-02

CONDITIONS: C-Section

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- immediate mother-skin-to-skin contact(SSC) (Experimental): The immediate mother-SSC begins directly after birth (still during the C-section)
  Interventions: Other: Skin-to-skin contact
- immediate father-SSC (Active Comparator): The immediate father-SSC begins directly after birth (still during C-section)
  Interventions: Other: Skin-to-skin contact
- Routine care;mother-SSC after 30 minutes (Other): After birth (still during C-section) the newborn gets routine care of a midwife close to the mother. SSC with mother after 30 minutes
  Interventions: Other: Skin-to-skin contact

INTERVENTIONS:
Other: Skin-to-skin contact

SUMMARY:
The randomised study analyzes the effects of immediate bonding (skin-to-skin contact) on different psychobiological and somatic outcomes of mother and child. The investigators compare 3 bonding conditions. Cortisol and Oxytocin are also measured during the bonding process.

ELIGIBILITY:
Inclusion Criteria:

* Mothers with elective Caesarean Section and their partners

Exclusion Criteria:

* premature birth
* severe diseases
* drug abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Changes in Cortisol Level | 30 and 60 minutes after bonding
  Cortisol is assessed as a stress parameter by Saliva. It will be tested in the mother and child to measure the effect of immediate bonding with the mother compared to the other 2 conditions on the stress level

SECONDARY OUTCOMES:
Depression | 1-3 days and 6 weeks after childbirth
  assessed by EPDS
Mother-child-bonding | 1-3 days and 6 weeks after childbirth
  assessed by PBQ
Child's heart ratio | 30 and 60 minutes after birth
Child's oxygen saturation | 30 and 60 minutes after birth
Child's temperature | 30 and 60 minutes after birth
Oxytocin | 30 and 60 minutes after birth
  Saliva measurement

CONTACTS AND LOCATIONS:
Overall Officials: Frank Louwen, Prof., Study Director — University Hospital Frankfurt-Dept. Obstetrics and Perinatal Medicine
Locations (1):
- University Hospital Frankfurt-Dept.Obstetrics and Perinatal Medicine, Frankfurt am Main, Hesse, Germany